CLINICAL TRIAL: NCT00951418
Title: Serum Clozapine and Cognition
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 1.5-15 July 2008
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-08

CONDITIONS: Schizophrenia
Keywords: clozapine; schizophrenia; cognition; t-wave morphology
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aim to investigate the relationship between serum levels of clozapine and cognitive performance in patients with ICD-10 Schizophrenia and treated with clozapine monotherapy. The hypothesis is that higher serum levels of clozapine are associated with cognitive dysfunctions. Furthermore, ECG changes and the relation to serum level of clozapine are studied. The design is cross-sectional.

ELIGIBILITY:
Inclusion Criteria:

* Treated with clozapine for minimum 6 months.
* Fixed dosage of clozapine last month before inclusion.

Exclusion Criteria:

* Substance misuse.
* Depression (Calgary Depression score ≥7).
* Somatic disease that interfere with cognitive performance.
* Treatment with benzodiazepines (half-lives >15 hours not allowed up 14 days prior inclusion and during study. Half-lives < 15 hours not allowed 3 days prior cognitive testing).
* Electroconvulsive therapy.
* Treatment with other antipsychotics.
* Withdrawal of informed consent.
* Compulsory measures.
* Treatment with anticholinergics except for atropine drops administered sublingually.
* Changes in use of tobacco last month before inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICD-10 Schizophrenia (f20.0-3; F20.9) treated with clozapine
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Cognitive function measured by CANTAB | once

SECONDARY OUTCOMES:
T-wave morphology | Once
Sedation VAS,ACES and SWAI scale | once

CONTACTS AND LOCATIONS:
Overall Officials: Rene Ernst Nielsen, M.D., Principal Investigator — Aalborg Psychiatric Hospital
Locations (1):
- Aalborg Psychiatric Hospital, Aalborg, Denmark